CLINICAL TRIAL: NCT04287543
Title: Effect of Melatonin Administration on the PER1 and BMAL1 Clock Genes in Patients With Parkinson's Disease
Brief Title: Melatonin on Clock Genes in Parkinson's Disease
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, we were unable to begin the study
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Blanca Miriam de Guadalupe Torres Mendoza, Head of aging laboratory, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2018-785-019
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease
Keywords: melatonin; clock genes; BMAL1 gene; PER1 gene
MeSH Terms: conditions — Parkinson Disease | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Experimental): Patients with PD who will receive 25 mg of melatonin gel at 12 hours a day and half an hour before sleeping for 12 months
  Interventions: Drug: Melatonin
- Placebo group (Placebo Comparator): Patients with PD who will receive 25 mg of placebo gel at 12 hours a day and half an hour before sleeping for 12 months
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Melatonin — 25 mg of melatonin gel at noon and 25 mg of melatonin gel 30 minutes before sleeping for 12 months
  Arms: Melatonin group
Drug: Placebos — 25 mg of placebo gel at noon and 25 mg of placebo gel 30 minutes before sleeping for 12 months
  Arms: Placebo group

SUMMARY:
Parkinson's disease (PD) is the second most important neurodegenerative disease that affects about 2% of the population over 60 years of age. About 40% of the Mexican population with PD suffer from sleep disorders, which has been linked to a deregulation of the circadian cycle and therefore of the clock genes. Melatonin is a hormone produced by the pineal gland that regulates the sleep-wake cycle, at pharmacological doses, it is used to decrease sleep disorders; it is suggested that is used could also normalize the levels of the clock genes expression. In rats with PD, a decrease in clock genes levels has been observed, which are restored by administering melatonin. The aim of the study is to evaluate the effect of melatonin on the expression of the PER1 and BMAL1 clock genes in patients with PD during 12 months. A controlled, double-blind, randomized clinical trial will be carried out in patients with a diagnosis of PD. A survey will be applied in order to know the course of the disease and two more tests to rule out some sleep disorder, at the beginning of the study, at the 6th month and at the 12th month. A blood sample (approximately 15 ml) will be taken every 3 months for a year. By random assignment, the participant will be given Melatonin or placebo, which should be taken every day in the morning and evening after meals for one year.

DETAILED DESCRIPTION:
A controlled, double-blind, randomized clinical trial will be carried out in 58 patients with a diagnosis of PD. Twenty-nine patients will receive Melatonin and 29 placebo. A blood sample will be taken to determine the expression levels of the PER1 and BMAL1 clock genes by a real-time quantitative polymerase chain reaction (RT-qPCR), and as secondary variables, to determine the activity of the mitochondrial complex 1, the levels of malondialdehyde (MDA) and 4-hydroxyalkene (4-HDA) and the production of nitric oxide will be quantified by spectrophotometric methods. The SCOPA-Sleep and EPWORTH questionnaires will be applied to assess sleep. To evaluate the clinical evolution of PD in each patient, the UPDRS scale will be used. It will be given the assigned treatment, with the printed patient code. They will be supplemented with 50 mg of Melatonin at a dose of 25 mg orally every 12 hours for 12 months. The double-blind of the medication for this study will be maintained by the use of gels identical to the Melatonin supplement. The blind's break will only be authorized in case of emergency events that require it, and the date, time and reason for the break should be noted. It will be given a follow-up diary, and the patient will be explained how they should take the treatment and that they should record the date and time of administration, the description of adverse events that may occur, raising the patient's awareness that It is important to keep the diary and take it at each appointment to assess the attachment to treatment. Concerning the medications that patients ingest, before entering the protocol, it will be indicated to follow their usual administration. Finally, the patient will be instructed to schedule their appointment 3,6, 9 and 12 months later of starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of PD in stages 1-3 of the classification by stages of Hoehn & Yahr
* Go with a companion to the appointments
* Patients who agree to participate in the study and sign the Informed Consent letter

Exclusion Criteria:

* Patients with movement disorder other than PD
* Prior pallidotomy, thalamotomy or deep brain stimulation
* Pregnant
* Patients who consume alcohol or coffee
* Patients who consume an antioxidant supplement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Expression levels of clock genes | Change from baseline at third, sixth, ninth and twelfth month
  Relative ratio of messenger ribonucleic acid (mRNA) expression of PER1 and BMAL1 genes corresponding to a control (GAPDH) for each sample, measured by an RT-qPCR.

SECONDARY OUTCOMES:
SCOPA-Sleep scale | Change from baseline at third, sixth, ninth and twelfth month
  It is a specific instrument for the evaluation of sleep disorders in patients with PD. It is self-applicable and consists of two subscales; the first assess nighttime sleep and the second daytime sleepiness during the last month. The score greater than seven of five points respectively indicates abnormal sleepiness. Additionally, the SCOPA-Sleep scale has a question of global sleep evaluation.
Epworth scale | Change from baseline at third, sixth, ninth and twelfth month
  Is an eight-item self-applicable instrument developed to assess the propensity to fall asleep in eight situations, mostly monotonous. A total score of less than 10 was considered normal, 10-12 as indicative of marginal drowsiness and above 12 suggestive of excessive drowsiness.
Progression of PD | Change from baseline at third, sixth, ninth and twelfth month
  For the longitudinal follow-up of the PD course, the Unified Parkinson's Disease Rating Scale (UPDRS) will be applied through an interview. The scale is composed by four parts: mental, behavioral and mood; activities of daily living; motor evaluation; and motor complications. The scoring range is from 0 to 199, where "199" represents total disability and "0" without disability.
Anxiety | Change from baseline at third, sixth, ninth and twelfth month
  To assess the severity of a person's anxiety symptoms and discriminate between anxiety and depression symptoms the Beck anxiety inventory will be use.
  The rating is made through a likert scale of 0 to 3, where 0 means absence of the symptom and 3 maximum severity. The total score is obtained from the sum of the 21 reagents, 0 is the minimum and 63 is the maximum. In the Mexican population, a score of 0-5 points will be minimal anxiety, 6-15 mild anxiety, 16-30 moderate anxiety and 31-63 severe anxiety.
Depression | Change from baseline at third, sixth, ninth and twelfth month
  To evaluate the severity of depression symptoms the Beck's depression inventory will be use. The rating is made through a likert scale of 0 to 3, where 0 means absence of the symptom and 3 maximum severity. The total score is obtained from the sum of the 21 reagents, 0 is the minimum and 63 is the maximum. In the Mexican population, a score of 0-9 points will be considered normal, 10-16 mild depression, 17-29 moderate depression, and 30-63 severe depression.
Activity of the mitochondrial complex 1 | Change from baseline at third, sixth, ninth and twelfth month
  To measure the mitochondrial complex I, a spectrophotometric assay will be used, it measures the oxidation of rotenone-sensitive nicotinamide-adenine dinucleotide (NADH) at 340 nm in mitochondria-enriched fractions
Oxidative stress | Change from baseline at third, sixth, ninth and twelfth month
  Products of nitric oxide metabolism and products of lipoperoxidation such as malondialdehyde and 4-hydroxyalkene by spectrophotometry will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Blanca M. Torres, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
It is planned to inform the patient individually about their results; if the results are favorable it will be considered to apply them to the Clinical of Movement Disorders patients. All data will be published in an article.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Poewe W, Seppi K, Tanner CM, Halliday GM, Brundin P, Volkmann J, Schrag AE, Lang AE. Parkinson disease. Nat Rev Dis Primers. 2017 Mar 23;3:17013. doi: 10.1038/nrdp.2017.13. PMID 28332488
- [Background] Barzilai A, Melamed E. Molecular mechanisms of selective dopaminergic neuronal death in Parkinson's disease. Trends Mol Med. 2003 Mar;9(3):126-32. doi: 10.1016/s1471-4914(03)00020-0. PMID 12657434
- [Background] Shadrina MI, Slominsky PA, Limborska SA. Molecular mechanisms of pathogenesis of Parkinson's disease. Int Rev Cell Mol Biol. 2010;281:229-66. doi: 10.1016/S1937-6448(10)81006-8. PMID 20460187
- [Background] Chung S, Bohnen NI, Albin RL, Frey KA, Muller ML, Chervin RD. Insomnia and sleepiness in Parkinson disease: associations with symptoms and comorbidities. J Clin Sleep Med. 2013 Nov 15;9(11):1131-7. doi: 10.5664/jcsm.3150. PMID 24235893
- [Background] Breen DP, Vuono R, Nawarathna U, Fisher K, Shneerson JM, Reddy AB, Barker RA. Sleep and circadian rhythm regulation in early Parkinson disease. JAMA Neurol. 2014 May;71(5):589-595. doi: 10.1001/jamaneurol.2014.65. PMID 24687146
- [Background] Cai Y, Liu S, Sothern RB, Xu S, Chan P. Expression of clock genes Per1 and Bmal1 in total leukocytes in health and Parkinson's disease. Eur J Neurol. 2010 Apr;17(4):550-4. doi: 10.1111/j.1468-1331.2009.02848.x. Epub 2009 Nov 12. PMID 19912323
- [Background] Videnovic A, Willis GL. Circadian system - A novel diagnostic and therapeutic target in Parkinson's disease? Mov Disord. 2016 Mar;31(3):260-9. doi: 10.1002/mds.26509. Epub 2016 Jan 30. PMID 26826022
- [Background] Cardinali DP, Pagano ES, Scacchi Bernasconi PA, Reynoso R, Scacchi P. Melatonin and mitochondrial dysfunction in the central nervous system. Horm Behav. 2013 Feb;63(2):322-30. doi: 10.1016/j.yhbeh.2012.02.020. Epub 2012 Feb 25. PMID 22391273
- [Background] Videnovic A, Golombek D. Circadian Dysregulation in Parkinson's Disease. Neurobiol Sleep Circadian Rhythms. 2017 Jan;2:53-58. doi: 10.1016/j.nbscr.2016.11.001. Epub 2016 Nov 12. PMID 28713867
- [Background] Elbaz A, Carcaillon L, Kab S, Moisan F. Epidemiology of Parkinson's disease. Rev Neurol (Paris). 2016 Jan;172(1):14-26. doi: 10.1016/j.neurol.2015.09.012. Epub 2015 Dec 21. PMID 26718594
- [Background] Perfeito R, Cunha-Oliveira T, Rego AC. Reprint of: revisiting oxidative stress and mitochondrial dysfunction in the pathogenesis of Parkinson disease-resemblance to the effect of amphetamine drugs of abuse. Free Radic Biol Med. 2013 Sep;62:186-201. doi: 10.1016/j.freeradbiomed.2013.05.042. Epub 2013 Jun 3. PMID 23743292
- [Background] Abou-Sleiman PM, Muqit MM, Wood NW. Expanding insights of mitochondrial dysfunction in Parkinson's disease. Nat Rev Neurosci. 2006 Mar;7(3):207-19. doi: 10.1038/nrn1868. PMID 16495942
- [Background] Mattam U, Jagota A. Daily rhythms of serotonin metabolism and the expression of clock genes in suprachiasmatic nucleus of rotenone-induced Parkinson's disease male Wistar rat model and effect of melatonin administration. Biogerontology. 2015 Feb;16(1):109-23. doi: 10.1007/s10522-014-9541-0. Epub 2014 Nov 28. PMID 25430725
- [Background] Ortiz GG, Benitez-King GA, Rosales-Corral SA, Pacheco-Moises FP, Velazquez-Brizuela IE. Cellular and biochemical actions of melatonin which protect against free radicals: role in neurodegenerative disorders. Curr Neuropharmacol. 2008 Sep;6(3):203-14. doi: 10.2174/157015908785777201. PMID 19506721
- [Background] Ortiz GG, Pacheco-Moises FP, Gomez-Rodriguez VM, Gonzalez-Renovato ED, Torres-Sanchez ED, Ramirez-Anguiano AC. Fish oil, melatonin and vitamin E attenuates midbrain cyclooxygenase-2 activity and oxidative stress after the administration of 1-methyl-4-phenyl-1,2,3,6- tetrahydropyridine. Metab Brain Dis. 2013 Dec;28(4):705-9. doi: 10.1007/s11011-013-9416-0. Epub 2013 May 24. PMID 23703110
- [Background] Trotti LM, Bliwise DL. Treatment of the sleep disorders associated with Parkinson's disease. Neurotherapeutics. 2014 Jan;11(1):68-77. doi: 10.1007/s13311-013-0236-z. PMID 24272458
- [Background] Medeiros CA, Carvalhedo de Bruin PF, Lopes LA, Magalhaes MC, de Lourdes Seabra M, de Bruin VM. Effect of exogenous melatonin on sleep and motor dysfunction in Parkinson's disease. A randomized, double blind, placebo-controlled study. J Neurol. 2007 Apr;254(4):459-64. doi: 10.1007/s00415-006-0390-x. Epub 2007 Apr 3. PMID 17404779
- [Background] Videnovic A, Zee PC. Consequences of Circadian Disruption on Neurologic Health. Sleep Med Clin. 2015 Dec;10(4):469-80. doi: 10.1016/j.jsmc.2015.08.004. Epub 2015 Sep 26. PMID 26568123
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Jankovic J. An update on the treatment of Parkinson's disease. Mt Sinai J Med. 2006 Jul;73(4):682-9. PMID 16878274
- [Background] Fernandez HH. Updates in the medical management of Parkinson disease. Cleve Clin J Med. 2012 Jan;79(1):28-35. doi: 10.3949/ccjm.78gr.11005. PMID 22219231
- [Background] Bolitho SJ, Naismith SL, Rajaratnam SM, Grunstein RR, Hodges JR, Terpening Z, Rogers N, Lewis SJ. Disturbances in melatonin secretion and circadian sleep-wake regulation in Parkinson disease. Sleep Med. 2014 Mar;15(3):342-7. doi: 10.1016/j.sleep.2013.10.016. Epub 2014 Jan 21. PMID 24529544
- [Background] Zhang Y, Chen J, Qiu J, Li Y, Wang J, Jiao J. Intakes of fish and polyunsaturated fatty acids and mild-to-severe cognitive impairment risks: a dose-response meta-analysis of 21 cohort studies. Am J Clin Nutr. 2016 Feb;103(2):330-40. doi: 10.3945/ajcn.115.124081. Epub 2015 Dec 30. PMID 26718417
- [Background] Taghizadeh M, Tamtaji OR, Dadgostar E, Daneshvar Kakhaki R, Bahmani F, Abolhassani J, Aarabi MH, Kouchaki E, Memarzadeh MR, Asemi Z. The effects of omega-3 fatty acids and vitamin E co-supplementation on clinical and metabolic status in patients with Parkinson's disease: A randomized, double-blind, placebo-controlled trial. Neurochem Int. 2017 Sep;108:183-189. doi: 10.1016/j.neuint.2017.03.014. Epub 2017 Mar 22. PMID 28342967
- [Background] Mayo JC, Sainz RM, Tan DX, Antolin I, Rodriguez C, Reiter RJ. Melatonin and Parkinson's disease. Endocrine. 2005 Jul;27(2):169-78. doi: 10.1385/ENDO:27:2:169. PMID 16217130
- [Background] Reiter RJ, Korkmaz A, Paredes SD, Manchester LC, Tan DX. Melatonin reduces oxidative/nitrosative stress due to drugs, toxins, metals, and herbicides. Neuro Endocrinol Lett. 2008 Oct;29(5):609-13. PMID 18987585
- [Background] Castellani RJ, Nunomura A, Rolston RK, Moreira PI, Takeda A, Perry G, Smith MA. Sublethal RNA oxidation as a mechanism for neurodegenerative disease. Int J Mol Sci. 2008 May;9(5):789-806. doi: 10.3390/ijms9050789. Epub 2008 May 20. PMID 19325784
- [Background] Reiter RJ. Oxidative damage in the central nervous system: protection by melatonin. Prog Neurobiol. 1998 Oct;56(3):359-84. doi: 10.1016/s0301-0082(98)00052-5. PMID 9770244
- [Background] Korkmaz A, Reiter RJ, Topal T, Manchester LC, Oter S, Tan DX. Melatonin: an established antioxidant worthy of use in clinical trials. Mol Med. 2009 Jan-Feb;15(1-2):43-50. doi: 10.2119/molmed.2008.00117. Epub 2008 Nov 4. PMID 19011689
- [Background] Mack JM, Schamne MG, Sampaio TB, Pertile RA, Fernandes PA, Markus RP, Prediger RD. Melatoninergic System in Parkinson's Disease: From Neuroprotection to the Management of Motor and Nonmotor Symptoms. Oxid Med Cell Longev. 2016;2016:3472032. doi: 10.1155/2016/3472032. Epub 2016 Oct 18. PMID 27829983
- [Background] Panigel M. [Application of new methods to the anatomical study of the human and animal placenta]. Bull Assoc Anat (Nancy). 1989 Sep;73(222):47-53. No abstract available. French. PMID 2700075
- [Background] Hartter S, Nordmark A, Rose DM, Bertilsson L, Tybring G, Laine K. Effects of caffeine intake on the pharmacokinetics of melatonin, a probe drug for CYP1A2 activity. Br J Clin Pharmacol. 2003 Dec;56(6):679-82. doi: 10.1046/j.1365-2125.2003.01933.x. PMID 14616429
- [Background] Weishaupt JH, Bartels C, Polking E, Dietrich J, Rohde G, Poeggeler B, Mertens N, Sperling S, Bohn M, Huther G, Schneider A, Bach A, Siren AL, Hardeland R, Bahr M, Nave KA, Ehrenreich H. Reduced oxidative damage in ALS by high-dose enteral melatonin treatment. J Pineal Res. 2006 Nov;41(4):313-23. doi: 10.1111/j.1600-079X.2006.00377.x. PMID 17014688
- [Background] Anderson G, Seo M, Berk M, Carvalho AF, Maes M. Gut Permeability and Microbiota in Parkinson's Disease: Role of Depression, Tryptophan Catabolites, Oxidative and Nitrosative Stress and Melatonergic Pathways. Curr Pharm Des. 2016;22(40):6142-6151. doi: 10.2174/1381612822666160906161513. PMID 27604608
- [Background] Vural EM, van Munster BC, de Rooij SE. Optimal dosages for melatonin supplementation therapy in older adults: a systematic review of current literature. Drugs Aging. 2014 Jun;31(6):441-51. doi: 10.1007/s40266-014-0178-0. PMID 24802882
- [Background] Lewy AJ, Sack RL, Miller LS, Hoban TM. Antidepressant and circadian phase-shifting effects of light. Science. 1987 Jan 16;235(4786):352-4. doi: 10.1126/science.3798117.
- [Background] Belaid H, Adrien J, Karachi C, Hirsch EC, Francois C. Effect of melatonin on sleep disorders in a monkey model of Parkinson's disease. Sleep Med. 2015 Oct;16(10):1245-51. doi: 10.1016/j.sleep.2015.06.018. Epub 2015 Jul 14. PMID 26429753
- [Background] Innominato PF, Lim AS, Palesh O, Clemons M, Trudeau M, Eisen A, Wang C, Kiss A, Pritchard KI, Bjarnason GA. The effect of melatonin on sleep and quality of life in patients with advanced breast cancer. Support Care Cancer. 2016 Mar;24(3):1097-105. doi: 10.1007/s00520-015-2883-6. Epub 2015 Aug 11. PMID 26260726
- [Background] Ortiz GG, Morales-Sanchez EW, Pacheco-Moises FP, Jimenez-Gil FJ, Macias-Islas MA, Mireles-Ramirez MA, Gonzalez-Usigli H. [Effect of melatonin administration on cyclooxygenase-2 activity, serum levels of nitric oxide metabolites, lipoperoxides and glutathione peroxidase activity in patients with Parkinson's disease]. Gac Med Mex. 2017;153(Supl. 2):S72-S81. doi: 10.24875/GMM.M000008. Spanish. PMID 29099102
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- See also: INEGI — http://www3.inegi.org.mx/sistemas/temas/default.aspx?s=est&c=17484